CLINICAL TRIAL: NCT00971737
Title: A Randomized, Open-Label Comparative Study of Combination Therapy With Cyclophosphamide and an Allogeneic GM-CSF-secreting Breast Tumor Vaccine With or Without Trastuzumab for the Treatment of Metastatic Breast Cancer That Does NOT Over-express HER-2/Neu
Brief Title: Cyclophosphamide and Vaccine Therapy With or Without Trastuzumab in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J0947; P30CA006973 (NIH); JHOC-J0947; NA_00024527; GENENTECH-JHOC-J0947; CDR0000653173 (Other: other)
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Trastuzumab; Cyclophosphamide

ARMS (2):
- Cyclophosphamide and Vaccine only (Active Comparator): Patients receive cyclophosphamide IV over 30 minutes on day -1 and allogeneic GM-CSF-secreting breast cancer vaccine intradermally on day 0. Courses repeat every 4-6 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients then receive a fourth vaccination at 6-8 months.
  Interventions: Biological: allogeneic GM-CSF-secreting breast cancer vaccine; Drug: cyclophosphamide
- Cyclophosphamide, Vaccine and Trastuzumab (Experimental): Patients receive cyclophosphamide and the vaccine as in arm I and trastuzumab IV over 30-90 minutes on day -1. Courses repeat every 4-6 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients then receive a fourth vaccination at 6-8 months.
  Interventions: Biological: allogeneic GM-CSF-secreting breast cancer vaccine; Biological: trastuzumab; Drug: cyclophosphamide

INTERVENTIONS:
Biological: allogeneic GM-CSF-secreting breast cancer vaccine — Given intradermally
Biological: trastuzumab — Given IV
  Arms: Cyclophosphamide, Vaccine and Trastuzumab
Drug: cyclophosphamide — Given IV

SUMMARY:
RATIONALE: Vaccines made from gene-modified tumor cells may help the body build an effective immune response to kill tumor cells. Biological therapies, such as cyclophosphamide and trastuzumab, may increase the number of immune cells and make the immune response stronger. It is not yet known whether giving cyclophosphamide together with vaccine therapy is more effective with or without trastuzumab in treating patients with metastatic breast cancer.

PURPOSE: This randomized phase II trial is studying the side effects of giving cyclophosphamide together with vaccine therapy and to see how well it works compared with giving cyclophosphamide and vaccine therapy together with trastuzumab in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the safety of cyclophosphamide-modulated vaccination with vs without trastuzumab in patients with breast cancer that does not overexpress HER-2/neu.
* To compare the clinical benefit of cyclophosphamide-modulated vaccination with vs without trastuzumab in these patients.
* To measure HER-2/neu-specific CD4+ and CD8+ T-cell immunity by delayed-type hypersensitivity (DTH) and ELISPOT.
* To measure the pharmacodynamics of CD4+CD25+ regulatory T cells by flow cytometry.

Secondary

* To assess the impact of trastuzumab on immune priming in vivo by immunohistochemistry of vaccine-site biopsies at day +3 and day +7 of courses 1 and 3 on the two study arms, comparing cellular infiltrates to those seen in previous preclinical and clinical models.
* To measure hTERT-specific CD8+ T-cell immunity by ELISPOT.
* To characterize the peripheral-memory T-cell pool.

Tertiary

* To determine baseline and change in vaccine site-draining lymph node immunohistology and gene expression profile.
* To develop the tandem tetramer/CD107a cytotoxicity assay for HER-2/neu-specific CD8+ T cells.
* To measure novel T-cell responses induced by trastuzumab and cyclophosphamide-modulated vaccination.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cyclophosphamide IV over 30 minutes on day -1 and allogeneic GM-CSF-secreting breast cancer vaccine intradermally on day 0. Courses repeat every 4-6 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients then receive a fourth vaccination at 6-8 months.
* Arm II: Patients receive cyclophosphamide and the vaccine as in arm I and trastuzumab IV over 30-90 minutes on day -1. Courses repeat every 4-6 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients then receive a fourth vaccination at 6-8 months.

Skin punch and lymph node biopsies are collected at baseline and on days +3 and +7 of courses 1 and 3 for biomarker analysis.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Does not overexpress HER-2/neu, defined as FISH negative or 0, 1+, or 2+ by IHC
  * Stage IV disease
* Must not be eligible for therapy of known curative potential for metastatic breast cancer
* Measurable or evaluable disease
* Stable CNS disease allowed provided that it's adequately treated and not under active treatment
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-1
* ANC > 1,000/mm^3
* Platelets > 100,000/mm^3
* Serum bilirubin < 2.0 mg/dL (unless due to Gilbert syndrome)
* AST and ALT < 2 times upper limit of normal (ULN)
* Alkaline phosphatase < 5 times ULN
* Serum creatinine < 2.0 mg/dL
* Ejection fraction normal by MUGA OR ≥ 50% by echocardiogram
* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* Asthma or chronic obstructive pulmonary disease that does not require daily systemic corticosteroids allowed
* No prior or concurrent autoimmune disease requiring management with systemic immunosuppression, including any of the following:

  * Inflammatory bowel disease
  * Systemic vasculitis
  * Scleroderma
  * Psoriasis
  * Multiple sclerosis
  * Hemolytic anemia or immune-mediated thrombocytopenia
  * Rheumatoid arthritis
  * Systemic lupus erythematosus
  * Sjogren syndrome
  * Sarcoidosis
  * Other rheumatologic disease
* No other malignancies within the past 5 years, except carcinoma in situ of the cervix, superficial nonmelanoma skin cancer, superficial bladder cancer, or tamoxifen-related endometrial cancer that has been adequately treated
* No active major medical or psychosocial problems that could be complicated by study participation
* No symptomatic intrinsic lung disease or extensive tumor involvement of the lungs resulting in dyspnea at rest
* No uncontrolled medical problems
* No evidence of active acute or chronic infection
* No known severe hypersensitivity to trastuzumab, except mild to moderate infusion reactions that are easily managed and do not recur
* No allergy to corn

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 28 days since prior and no other concurrent chemotherapy, radiation therapy, or biologic therapy (except trastuzumab)

  * Concurrent endocrine therapy and supportive therapy with bisphosphonates allowed
* More than 28 days since prior and no other concurrent participation in an investigational new drug trial
* More than 28 days since prior and no other concurrent systemic oral steroids

  * Topical, ocular, and nasal steroids allowed
* No prior vaccination with the allogeneic GM-CSF-secreting breast tumor vaccine

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leisha A. Emens, MD, PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 subjects were withdrawn prior to receiving intervention (2 due to development of new medical problems, 1 due to anxiety and non-compliance).
Period: Overall Study
Arm/Group | Cyclophosphamide and Vaccine Only | Cyclophosphamide, Vaccine and Trastuzumab
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 63 subjects were deemed eligible for this study. 2 were taken off-study prior to vaccination due to the development of new medical problems. 1 subject was taken off due to anxiety and non-compliance. 60 research subjects went on to receive at least 1 vaccination, where 30 subjects were randomized to Arm A and 30 subjects were randomized to Arm B.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclophosphamide and Vaccine Only | Cyclophosphamide, Vaccine and Trastuzumab | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 25 | 52
  >=65 years | 3 | 5 | 8
Age, Continuous [Mean (Full Range); unit: years] | 53 [25 to 73] | 52 [34 to 69] | 53 [25 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Toxicity as Assessed by Number of Grade 3 or 4 Adverse Events
Description: Number of grade 3 or 4 nonhematologic toxicity (except alopecia), or any grade 4 hematologic toxicity as defined by NCI CTCAE v3.0
Time Frame: 3 years
Population: Data was not evaluable in 2/30 participants from the cyclophosphamide and vaccine-only arm.
Measure: Number; unit: adverse events
Arm/Group | Cyclophosphamide and Vaccine Only | Cyclophosphamide, Vaccine and Trastuzumab
Number analyzed (Participants) | 28 | 30
adverse events | 0 | 2

2. Primary Outcome: Clinical Benefit (CB) as Assessed by Progression Free Survival at Six Months
Description: Progression-free survival is measured as percentage of participants with stable disease or complete response, as defined by RECIST criteria, six months after receiving last vaccination. Progressive disease (PD) will be defined by the appearance of a new lesion, or by an increase of at least 20% in the sum of the longest diameter of target lesions, taking as a reference that smallest sum longest diameter recorded since the study intervention began. In the case of bone lesions, progressive disease will be established after eight weeks of increasing or new lesions if there is subjective progressive disease as noted by increasing bone pain or decreasing performance status. These observations must be present for at least two measurement periods separated by at least four weeks.
Time Frame: 6 months post-intervention
Population: Data was not evaluable in 2/30 participants from the cyclophosphamide and vaccine-only arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclophosphamide and Vaccine Only | Cyclophosphamide, Vaccine and Trastuzumab
Number analyzed (Participants) | 28 | 30
percentage of participants | 33 [17 to 53] | 37 [20 to 56]

3. Primary Outcome: HER-2/Neu-specific Immune Responses as Measured by Number of Participants With Positive for Delayed-type Hypersensitivity (DTH) Response
Time Frame: 3 years
Population: Data was not evaluable in 2/30 participants from the cyclophosphamide and vaccine-only arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide and Vaccine Only | Cyclophosphamide, Vaccine and Trastuzumab
Number analyzed (Participants) | 28 | 30
Participants | 14 | 16

4. Primary Outcome: Pharmacodynamics of Peripheral CD4+CD25+ Regulatory T Cells
Time Frame: 3 years
Population: Lab analysis could not be completed due to loss of funding, therefore data was not collected to assess this outcome measure.
Arm/Group | Cyclophosphamide and Vaccine Only | Cyclophosphamide, Vaccine and Trastuzumab
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Immune Priming in In-vivo Vaccine-site Biopsies
Time Frame: 3 years
Population: as for outcome 4
Arm/Group | Cyclophosphamide and Vaccine Only | Cyclophosphamide, Vaccine and Trastuzumab
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Enumeration of CD8+ T Cells Specific for hTERT by ELISPOT
Time Frame: 3 years
Population: as for outcome 4
Arm/Group | Cyclophosphamide and Vaccine Only | Cyclophosphamide, Vaccine and Trastuzumab
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Characterization of the T-cell Memory Pool Pre- and Post-vaccination
Time Frame: 3 years
Population: as for outcome 4
Arm/Group | Cyclophosphamide and Vaccine Only | Cyclophosphamide, Vaccine and Trastuzumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 6 months post-intervention
Arm/Group | Cyclophosphamide and Vaccine Only | Cyclophosphamide, Vaccine and Trastuzumab
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 30/30 | 30/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide and Vaccine Only (N=30) | Cyclophosphamide, Vaccine and Trastuzumab (N=30)
Erythema/swelling of vaccine sites (Skin and subcutaneous tissue disorders) | 30 (82) | 30 (102)
Pain/soreness/tenderness of vaccine sites (Skin and subcutaneous tissue disorders) | 28 (81) | 30 (82)
Pruritus of vaccine sites (Skin and subcutaneous tissue disorders) | 30 (78) | 30 (92)
Rash around vaccine sites (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3)
Blister at vaccine site (Skin and subcutaneous tissue disorders) | 16 (28) | 20 (41)
Ecchymosis at vaccine site (Skin and subcutaneous tissue disorders) | 8 (10) | 18 (24)
Hyperpigmentation at vaccine site (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Warmth at vaccine site (Skin and subcutaneous tissue disorders) | 16 (26) | 17 (34)
Anorexia (Gastrointestinal disorders) | 13 (22) | 10 (17)
Aphthus Ulcers (Gastrointestinal disorders) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (32) | 19 (33)
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 16 (29) | 15 (27)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dermatographism (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dry throat (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 3 (5) | 2 (3)
Fatigue (General disorders) | 16 (34) | 18 (32)
Fever (General disorders) | 11 (18) | 11 (17)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flu-like symptoms (General disorders) | 2 (2) | 2 (3)
Headache (Nervous system disorders) | 11 (21) | 15 (18)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection, Herpes (Infections and infestations) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 2 (5) | 6 (8)
Lymphadenopathy (Blood and lymphatic system disorders) | 9 (14) | 19 (31)
Malaise (General disorders) | 2 (2) | 3 (4)
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 16 (41) | 22 (37)
Nausea (Gastrointestinal disorders) | 12 (16) | 8 (10)
Neck stiffness (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Pain, bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain, hip/groin (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 7 (10) | 9 (12)
Sweats (General disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (4) | 5 (5)
Vaccine flare (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (3)
Hives (Skin and subcutaneous tissue disorders) | 2 (9) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes